CLINICAL TRIAL: NCT06742580
Title: The Relationship Between Idiopathic Acute Peripheral Facial Paralysis and Homocysteine Level in Adult Patients
Status: Recruiting | Type: Observational
Sponsor: Murat Akın (Other)
Responsible Party: Sponsor-Investigator, Murat Akın, assistant doctor, Afyonkarahisar Health Sciences University
Organization: Afyonkarahisar Health Sciences University (Other)
Other Study IDs: AFSÜ-KBB-MA-01
Record Dates: First submitted 2024-12-13; First posted 2024-12-19 (Actual); Last update posted 2024-12-19 (Actual); Status verified 2024-12

CONDITIONS: Facial Paralysis, Peripheral; Bell Palsy
Keywords: Acute Peripheral Facial Paralysis; Homocysteine; Bell Palsy
MeSH Terms: conditions — Facial Paralysis; Bell Palsy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Bell palsy patient group: Patients who applied to our hospital due to idiopathic facial paralysis within the first month
- control group: Healthy individuals with no known health problems

SUMMARY:
In the etıology of Idıopathıc Acute Perıpheral Facıal Palsy, known as bell palsy, many causes have been descrıbed, such as specıfıc ımmune, ıchemıc, ınfectıous and heredıal factors. ın our study, we have observed the blood homocysteıne level that causes thrombotıc dısorders ın paralysıs patıents.

DETAILED DESCRIPTION:
Bell's palsy, also known as "acute facial palsy of unknown cause", is a common cranial neuropathy that characteristically causes facial muscle paresis or complete paralysis on one side, occurs suddenly and may progress over 48 hours. It is accompanied by postauricular pain, dysgeusia, subjective alteration of facial sensation, and hyperacusis. Bell's palsy accounts for 60-75 percent of all cases of facial palsy. It occurs in 7-40 cases per 100,000 people each year, and the prevalence is similar in both sexes. Its cause remains idiopathic, but it is strongly associated with certain viral infections, which cause neuritis leading to focal edema, demyelination, and ischemia. Although the exact pathogenesis of Bell's palsy is unknown and is considered idiopathic, specific immune, ischemic, and hereditary factors are strongly associated with its etiology. Homocysteine is an amino acid that is not provided by the diet and can be converted to cysteine with the help of specific B vitamins or converted back to methionine, an essential amino acid. Homocysteine levels vary between men and women and are usually in the normal range of 5 to 15 micromoles/L. When homocysteine levels exceed 15 micromoles/L, it is called hyperhomocysteinemia.

The estimated prevalence of mild hyperhomocysteinemia in the general population is 5% to 7%. Several studies have shown that it is an independent risk factor for thrombotic disorders (i.e., deep vein thrombosis). It has even been reported that lowering a patient's homocysteine level by 25% reduces the risk of stroke by 19%.

A significant relationship was found in the meta-analysis conducted in the literature regarding sudden sensorineural hearing loss and high homocysteine levels. Due to the similar anatomical location of the facial nerve and N. vestibulocochlearis, it was planned to examine the relationship between acute idiopathic peripheral paralysis and homocysteine. There is no previous study in the literature. Therefore, this study will be the pioneering research in the literature regarding blood homocysteine levels in patients diagnosed with Idiopathic Acute Peripheral Facial Paralysis.

ELIGIBILITY:
Inclusion Criteria:

- Patients admitted with acute facial paralysis

Exclusion Criteria:

* Facial and ear trauma or tumor
* İatrogenic
* Cholesteatoma
* Facial paralysis due to central nervous system diseases

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: AFYON HEALTH SCIENCES UNIVERSITY HOSPITAL
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-08-04 (Estimated)

PRIMARY OUTCOMES:
Homosystein test results | up to 24 weeks
  The results have not been obtained from lab yet. So none results were measured .

CONTACTS AND LOCATIONS:
Overall Officials: Orhan Kemal KAHVECİ, PROFESSOR, Principal Investigator — AFYON HEALTH SCIENCES UNIVERSITY HOSPITAL
Locations (1):
- Afyonkarahisar Health Sciences University, Afyonkarahisar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
WILL BE DECLARED AT THE RESULT OF THE STUDY

REFERENCES:
- [Background] Singh A, Deshmukh P. Bell's Palsy: A Review. Cureus. 2022 Oct 11;14(10):e30186. doi: 10.7759/cureus.30186. eCollection 2022 Oct. PMID 36397921
- [Background] Son P, Lewis L. Hyperhomocysteinemia. 2022 May 8. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK554408/ PMID 32119295
- [Background] Niu X, Chen Y, Zhong Y, Xiao X. The relationship between serum homocysteine levels and sudden sensorineural hearing loss: a meta-analysis. Eur Arch Otorhinolaryngol. 2023 May;280(5):2091-2097. doi: 10.1007/s00405-023-07829-w. Epub 2023 Jan 19. PMID 36658368
- [Background] Eviston TJ, Croxson GR, Kennedy PG, Hadlock T, Krishnan AV. Bell's palsy: aetiology, clinical features and multidisciplinary care. J Neurol Neurosurg Psychiatry. 2015 Dec;86(12):1356-61. doi: 10.1136/jnnp-2014-309563. Epub 2015 Apr 9. PMID 25857657